CLINICAL TRIAL: NCT01680913
Title: Does Ultrasound Guidance Improve Time to Perform a Spinal or Number of Attempts in Obese Patients? A Randomized Controlled Study.
Brief Title: Does Ultrasound Guidance Improve Time to Perform a Spinal or Number of Attempts in Obese Patients?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Jacelyn Larson, Faculty, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: U/S spinals
Record Dates: First submitted 2012-08-28; First posted 2012-09-07 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Spinal Anesthesia Administration
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spinal with ultrasound guidance (Experimental): The intervention group's interspaces will be determined using the curved linear probe on a Zonare ultrasound using two views.
  Interventions: Procedure: Ultrasound guidance; Procedure: Spinal anesthetic
- Spinal by palpation of Tuffier's line (Active Comparator): Current clinical practice. Standard of care would have the attending anesthetist palpate the Tuffier's line to pinpoint the appropriate location for the spinal.
  Interventions: Procedure: Palpation of Tuffier's line; Procedure: Spinal anesthetic

INTERVENTIONS:
Procedure: Ultrasound guidance — The intervention group's interspaces will be determined using the curved linear probe on a Zonare ultrasound using two views.
  Arms: Spinal with ultrasound guidance
Procedure: Palpation of Tuffier's line — Current clinical practice. Standard of care would have the attending anesthetist palpate the Tuffier's line to pinpoint the appropriate location for the spinal.
  Arms: Spinal by palpation of Tuffier's line
Procedure: Spinal anesthetic — Subcutaneous local infiltration with a 25g needle we be performed prior to the spinal. Neuraxial technique will be attempted midline with a 25 gauge whitacre needle in the sitting position. Spinals will be attempted on either L2-L3, L3-L4, L4-L5 interspaces. The amount and type of local anesthetic/intrathecal narcotic will be left to the discretion of the Anesthetist.

SUMMARY:
Spinal anesthesia depends on being able to locate physical landmarks on a patient's body. In obese patients, the commonly used landmarks may be difficult or even impossible to feel. In addition, the spine can be hidden beneath a layer of fatty tissue.

Ultrasound is useful for finding the correct injection site in pregnant patients, but the usefulness of ultrasound has not been adequately evaluated in non-pregnant patients. The potential benefits for obese patients from the use of ultrasound include shortening the duration of the procedure, increasing patient comfort, decreasing the total number of attempts, and aiding in the choice of appropriate needle length for the patient.

The investigators hypothesize that there is no difference in time to perform a spinal anesthetic when landmarking with ultrasound as compared to tactile landmarking in patients with BMI > 35.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgeries amenable to spinal anesthetic
* BMI >35
* between the ages of 18-85

Exclusion Criteria:

* Patients with known spinal disease or previous spinal surgery
* Pregnant patients
* Patients requiring emergent surgeries
* Patients in positions other than sitting during neuroaxial anesthesia
* Patients with contraindications to neuroaxial anesthesia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Total time to perform the spinal | From the beginning of palpation or ultrasound to free flow of Cerebral Spinal Fluid (CSF), up to 1 hour.

SECONDARY OUTCOMES:
Time from administration of the local anesthetic needle until free flow CSF | Up to 1 hour
Number of needle redirections | At time of spinal anesthetic administration
Number of attempts to complete the spinal | At time of spinal anesthetic administration
  As measured by new needle puncture sites, according to the anesthetist performing the procedure
Number of failed blocks | Up to 15 minutes after administration of spinal anesthesia
  Defined as unable to get free flow CSF or inadequate surgical block after administration of neuraxial anesthetic after 15 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Jacelyn Larson, MD FRCP, Principal Investigator — University of Saskatchewan
Locations (2):
- Canada (2):
  - Saskatoon City Hospital, Saskatoon, Saskatchewan
  - Saint Paul's Hospital, Saskatoon, Saskatchewan